CLINICAL TRIAL: NCT02574988
Title: The Multicenter Registry of Patients With Severe Cutaneous Adverse Reactions Among Tertiary Medical Institutes in Thailand
Brief Title: Severe Cutaneous Adverse Reactions in Thailand
Acronym: ThaiSCAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Chiang Mai University (Other); Thammasat University (Other); Phramongkutklao College of Medicine and Hospital (Other); Mahidol University (Other)
Responsible Party: Principal Investigator, Jettanong Klaewsongkram, Jettanong Klaewsongkram, MD., Chulalongkorn University
Other Study IDs: Chula-ARC 001/15
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Steven-Johnson Syndrome; Toxic Epidermal Necrolysis; Drug Reaction With Eosinophilia and Systemic Symptoms; Acute Generalized Exanthematous Pustulosis; Generalized Bullous Fixed Drug Eruption
Keywords: drug allergy; drug hypersensitivity; adverse drug reactions; severe cutaneous adverse reactions
MeSH Terms: conditions — Stevens-Johnson Syndrome; Drug Hypersensitivity Syndrome; Acute Generalized Exanthematous Pustulosis; Drug Hypersensitivity; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — cryopreserved peripheral blood mononuclear cells, buffy coat, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SCAR Patients: Patients diagnosed with severe cutaneous adverse reactions with be recruited

SUMMARY:
The multicenter registry of patients with severe cutaneous adverse reactions among tertiary medical institutes in Thailand to study clinical characteristics, etiologies, therapeutic outcomes, quality of life, and the values of in vitro drug allergy diagnosis for the confirmation of the causative drugs

DETAILED DESCRIPTION:
Patients with severe cutaneous adverse reactions (Steven-Johnson Syndrome, toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms, acute generalized exanthematous pustulosis, and generalized bullous fixed drug eruption) among six tertiary medical institutes in Thailand will be recruited to study clinical characteristics, etiologies, therapeutic outcomes, quality of life, and the values of using laboratory techniques for the confirmation of the causative drugs

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled criteria of probable or definite cases of SJS, TEN, DRESS, or AGEP according to RegiSCAR validation criteria as well as patients diagnosed with GBFDE

Exclusion Criteria:

* Patients later confirmed to have other diagnosis than diseases mentioned above or have no sufficient data for the registry

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), drug reaction with eosinophilia and systemic symptoms (DRESS), acute generalized exanthematous pustulosis (AGEP), or generalized bullous fixed drug eruption (GBFDE) from 6 tertiary medical centers in Thailand with be recruited into this registry
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 1 year
Diagnostic values of in vitro tests for drug allergy diagnosis | 1 year

SECONDARY OUTCOMES:
Complications | 1 year
  Percentages of patients suffer from severe cutaneous adverse reactions will be reported and categorized according to organ involvement
Quality of Life | 1 year
  Patient's quality of life will be assessed by using The World Health Organization Quality of Life (WHOQOL)-BREF; Thai version and The Drug Hypersensitivity Quality of Life Questionnaire (DrHy-Q); Thai version

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klaewsongkram J, Sukasem C, Thantiworasit P, Suthumchai N, Rerknimitr P, Tuchinda P, Chularojanamontri L, Srinoulprasert Y, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C; ThaiSCAR study group. Analysis of HLA-B Allelic Variation and IFN-gamma ELISpot Responses in Patients with Severe Cutaneous Adverse Reactions Associated with Drugs. J Allergy Clin Immunol Pract. 2019 Jan;7(1):219-227.e4. doi: 10.1016/j.jaip.2018.05.004. Epub 2018 May 22. PMID 29800753
- [Result] Suthumchai N, Srinoulprasert Y, Thantiworasit P, Rerknimitr P, Tuchinda P, Chularojanamontri L, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C, Sukasem C, Klaewsongkram J; ThaiSCAR study group. The measurement of drug-induced interferon gamma-releasing cells and lymphocyte proliferation in severe cutaneous adverse reactions. J Eur Acad Dermatol Venereol. 2018 Jun;32(6):992-998. doi: 10.1111/jdv.14890. Epub 2018 Mar 13. PMID 29478292
- [Result] Klaewsongkram J, Thantiworasit P, Suthumchai N, Rerknimitr P, Sukasem C, Tuchinda P, Chularojanamontri L, Srinoulprasert Y, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C. In vitro test to confirm diagnosis of allopurinol-induced severe cutaneous adverse reactions. Br J Dermatol. 2016 Nov;175(5):994-1002. doi: 10.1111/bjd.14701. Epub 2016 Aug 29. PMID 27106261
- [Result] Chongpison Y, Rerknimitr P, Hurst C, Mongkolpathumrat P, Palapinyo S, Chularojanamontri L, Srinoulprasert Y, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C, Sukasem C, Tuchinda P, Baiardini I, Klaewsongkram J. Reliability and validity of the Thai Drug Hypersensitivity Quality of Life Questionnaire: a multi-center study. Int J Qual Health Care. 2019 Aug 1;31(7):527-534. doi: 10.1093/intqhc/mzy207. PMID 30346532
- [Derived] Chongpison Y, Sriswasdi S, Buranapraditkun S, Thantiworasit P, Rerknimitr P, Mongkolpathumrat P, Chularojanamontri L, Srinoulprasert Y, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C, Sukasem C, Tuchinda P, Pongcharoen P, Klaewsongkram J. IFN-gamma ELISpot-enabled machine learning for culprit drug identification in nonimmediate drug hypersensitivity. J Allergy Clin Immunol. 2024 Jan;153(1):193-202. doi: 10.1016/j.jaci.2023.08.026. Epub 2023 Sep 9. PMID 37678574
- [Derived] Klaewsongkram J, Buranapraditkun S, Thantiworasit P, Rerknimitr P, Tuchinda P, Chularojanamontri L, Rerkpattanapipat T, Chanprapaph K, Disphanurat W, Chakkavittumrong P, Tovanabutra N, Srisuttiyakorn C, Srinoulprasert Y, Sukasem C, Chongpison Y. The Role of In Vitro Detection of Drug-Specific Mediator-Releasing Cells to Diagnose Different Phenotypes of Severe Cutaneous Adverse Reactions. Allergy Asthma Immunol Res. 2021 Nov;13(6):896-907. doi: 10.4168/aair.2021.13.6.896. PMID 34734507